CLINICAL TRIAL: NCT03254524
Title: Statewide Analysis of Emergency Department Use for Determining Geographic Patterns of Emergency Care Use, Hospital Choice and Measures of Population Health.
Brief Title: Geography of ED Use and Population Health
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01408
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Emergencies; Diabetes Mellitus
Keywords: Epidemiology Research
MeSH Terms: conditions — Emergencies; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients visiting an emergency department in New York State
  Interventions: Other: Statewide Planning and Research Cooperative System Database

INTERVENTIONS:
Other: Statewide Planning and Research Cooperative System Database — The Statewide Planning and Research Cooperative System (SPARCS) is a comprehensive data reporting system created to collect information on discharges from hospitals. SPARCS currently collects patient level detail on patient characteristics, diagnoses and treatments, services, and charges for every hospital discharge, ambulatory surgery patient, and emergency department admission in New York State.
  Other Names: SPARCS

SUMMARY:
The goal of this study is to create predictive models of emergency care and metrics for population health that can be used to analyze how events like hospital closures or disasters like Hurricane Sandy affect health care utilization by patients in specific populations or geographic regions. Additionally, it will allow the development of metrics for population health that can act as surveillance mechanisms to measure disease prevalence and identify patterns in emergency department use that can be used to identify specific geographic regions where health care is either optimized to promote health or needs to be improve so that population health can be improved.

DETAILED DESCRIPTION:
The purpose of this study is to analyze the geographic patterns of emergency department utilization. This study will look at the relationship that geographic proximity and local population factors have on patient use of emergency departments. Geographic proximity of alternative hospitals and elicit other patient and hospital specific factors, such as demographic, insurance type, diagnosis, and socioeconomic factors that lead patients to choose specific hospitals for emergency care or generally lead to patients accessing emergency care will be compared.

Patterns of emergency department utilization by patients will be identified in specific geographies such as Census tracts to determine clusters of high and low emergency department use. We also analyze the patterns of emergency care use based on specific disease conditions.Investigators will analyze the rate of emergency department use for patients with diabetes to determine population prevalence of diseases using emergency department data. Studying the pattern of use by specific geographies or disease conditions will also allow us to understand how emergency department use varies among populations by geographies and the socioeconomic and health care factors local to those regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting an emergency department in New York State

Exclusion Criteria:

* Depending on the population analyzed, may exclude some subpopulations such as children (in order study adults), prisoners or patients transferred from other healthcare facilities (in order to study non-institutionalized individuals).

Max Age: 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Includes all patients visiting an emergency department in New York State
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Emergency Deparrtment (ED) visit by a patient | 1 Day
  In order to identify repeat ED visits by the same individual, unique identifiers within SPARCS match visits by the same individual throughout the study period

SECONDARY OUTCOMES:
Surveillance of Disease Prevalence | 1 Day
  Proportion of individuals who recieve a given diagnosis like diabetes during any emergency department visit including emergency inpatient admissions.
Extension to Other Disease Conditions and Geographies | 1 Day
  Analysis of how disease prevalence can be measured at the level of the entire state. Populations will be stratified based on geography.
Hospital Selection | 1 Day
  Identification of the selection of a given hospital by patients based on facility codes contained within the SPARCS database.

CONTACTS AND LOCATIONS:
Overall Officials: David Lee, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States